CLINICAL TRIAL: NCT04272450
Title: Respiratory Muscle Strength in Different Age Groups_Turkey
Brief Title: Respiratory Muscle Strength in Different Age Groups
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal investigator, Istanbul Medipol University Hospital
Other Study IDs: MIPMEP_Turkey
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2022-11

CONDITIONS: Healthy Adults
Keywords: respiratory muscle; mouth pressure; normative data; predicted value; respiratory muscle strenght; Turkey; Istanbul

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: respiratory muscle strenght measurement — Maximum inspiratory pressure-maximum expiratory pressure. The mouth pressure measurement was performed with the Micro-RPM® instrument from SensorMEDIC. Patient placed a rubber mouthpiece with flanges, on the device, sealed their lips firmly around the mouthpiece, exhaled/inhaled slowly and completely and then tried to breath in as hard as possible. The patient was allowed to rest for about a minute and the maneuver was repeated.

SUMMARY:
In determining respiratory muscle strength, mouth pressure measurement is most frequently used in the clinic. Determination of respiratory muscle strength loss provides benefits such as taking the decision to use individual rehabilitation methods, making the decision for extubation in patients with mechanical ventilation. But Turkey normative values, these values are not available. In the investigator's country, the respiratory muscle forces of the cases are evaluated by comparing them with the normal / expected values of the Scandinavian races that do not have similar anatomical features with the Turkish society, which causes errors in diagnosis.

The 250 healthy cases, whose age ranges are between 20-70, 20-29, 30-40, 40-49, 50-59 and 60-70, will be examined by a pulmonologist and asked if they have any disease that may affect respiratory muscle strength. Mouth pressure measurements will be made for healthy and inclusion criteria, and maximal inspiratory and expiratory pressure distributions will be examined.

ELIGIBILITY:
Inclusion Criteria:

* The age range is 20-70,
* Body mass index to be 18.0- 29.5 kg / m2
* No cardiac, neuromuscular or endocrine disease that may affect any respiratory muscle strength Respiratory function parameters to be normal,
* Not being a smoker

Exclusion Criteria:

* Not agreeing to participate in the study
* Not being able to adapt to the device

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strenght measurement | 30 minutes
  Respiratory mus cle strength will be measured by measuring mouth pressure. Maximal inspiratory (MIP) and expiratory pressures (MEP) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided